CLINICAL TRIAL: NCT06613451
Title: The Effect of Mobile Application Use on the Intravenous, Intramuscular and Subcutaneous Drug Administration Knowledge and Skill Level of Pediatric Nursing Students: Randomized Controlled Study
Brief Title: The Effect of Mobile Application Use on Drug Administration Knowledge and Skill Level of Pediatric Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Rukiye Çelik, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1919B012312024
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Nurse's Role; Nursing Caries
Keywords: nurse student; RCT; drug administration; mobile application

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Care Provider
Masking Description: Nursing Student
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Mobil application
  Interventions: Other: Mobile Application
- Control Group (Active Comparator): standard undergraduate education
  Interventions: Other: Mobile Application

INTERVENTIONS:
Other: Mobile Application — Mobile Application Use on the Intravenous, Intramuscular and Subcutaneous Drug Administration

SUMMARY:
Care forms the basis of the nursing profession. Nurses have many roles, duties and responsibilities in the care process. One of these roles is safe drug practices within the scope of its therapeutic/healing role. Safe medication practices are an important component of patient safety, which is one of the most important indicators of quality in health care services. The pediatric patient group is a group at risk for medication errors. The reasons for this situation include the developmental characteristics of the pediatric group, their anatomical differences, their bioavailability, pharmacokinetic properties and pharmacodynamic properties compared to adults, the lack of ready-made forms of pediatric dose drugs, the excess of nurses' care practices in pediatric children, the limited communication ability of the pediatric patient, lack of personnel, medication for the pediatric group. There are deficiencies in application knowledge and skills. Medication errors can lead to fatal situations for children. There are a number of improvements made to prevent this situation. Despite all the improvements, it is seen that nurses continue to experience difficulties in drug preparation and administration, and medication administration is still a significant problem. One of the most important steps in solving this problem is the training on drug administration to be given during undergraduate education. Considering the learning skills and preferences of undergraduate nursing students living in adolescence, it is seen that they have a predisposition to technology, their ability to use it in daily life, and their interests. For this reason, it seems that technology-based applications can be used to help students learn medication practices more willingly, permanently and effectively. Technology and mobile applications; It is a learning method that affects all tactile, visual and kinesthetic areas. Use of technology in education; It develops independent learning skills, increases active learning, and offers different types of learning strategies together. It is planned to examine the effect of the mobile application developed with the planned project on the knowledge and skill level of intravenous (IV), intramuscular (IM) and subcutaneous (SC) drug applications, which are among the pediatric drug applications that are frequently mistaken in the literature.

DETAILED DESCRIPTION:
Care forms the basis of the nursing profession. Nurses have many roles, duties and responsibilities in the care process. One of these roles is the therapeutic/healing role. Its therapeutic/healing role has an important place in long and close relationships with healthy and sick individuals. In this role, one of the most important duties of nurses is safe medication administration. Safe medication practices are also an important component of patient safety, which is one of the most important indicators of quality in health care services. If the drug application in question is to be performed on a pediatric patient, pediatric characteristics should be known and awareness and more care should be taken. It has been reported that medication errors occur seven times more frequently in pediatric intensive care units than in other intensive care units. In a study, it was stated that 48.9% of nurses working in the field of pediatrics made a medication administration error at least once. The reasons for this situation include the developmental characteristics of the pediatric group, their anatomical differences, bioavailability, pharmacokinetic properties and pharmacodynamic properties compared to adults, the lack of ready-made forms of pediatric dose drugs, the need to adapt adult type drugs for children, the abundance of nurses' care practices in pediatric children, and the limited ability of the pediatric patient to communicate. , there is a lack of personnel and inadequacies in medication administration knowledge and skills for the pediatric group.

Although nurses have a very important impact on the diagnosis, treatment and prevention of diseases when medications are administered correctly, their incorrect administration can lead to many negative situations for the patient. In order for nurses to be able to administer medication in accordance with the principle of benefit / no harm, they need to have the ability to calculate drug dosage and master the techniques and steps of drug administration. In a study, in order to minimize all these application errors and ensure patient safety, equipment connected to information and automation technology, use of smart pump technology, patient wristbands, electronic prompts, use of electronic badges, patient tracking systems, and stocking with electronic barcoding are used during drug administration. Although the use of systems, PYXIS medication management system and a hospital information system integrated with all these systems has become widespread, it has been mentioned that nurses continue to experience difficulties in drug preparation and administration, and medication administration is still an important problem. One of the most important steps in solving this problem is the training on drug administration to be given during undergraduate education.

Nursing students are prone to making medical errors due to reasons such as not having completed their education yet and not starting to fully assume patient responsibility. Especially in drug applications that require extra attention and knowledge, and where even the slightest dose calculation and administration route error can cause sequelae and even fatal consequences, the undergraduate education that students will receive is important in preventing drug errors in clinical patient care in the future. However, it has been observed that students are inadequate in this regard and their calculation and application skills are not fully developed. A study supports this and emphasizes that senior nursing students fail 98% of dose calculation problems and that more practice should be done in mathematics and drug dose calculation during nursing education. For this reason, it is of great importance to provide practices to improve the knowledge and skills of nursing students regarding medication administration during their undergraduate education. However, studies show that the education given to nursing students is insufficient in terms of providing pharmacological knowledge and dose calculation skills in terms of patient safety. It has been observed that nursing students can make more observations about drug applications during their compulsory clinical training to improve their knowledge and skills, make calculations during the preparation of drugs, and have theoretical discussions with nurses and faculty members rather than practice in order to obtain the correct drug dose. In addition, considering the learning skills and preferences of undergraduate nursing students living in adolescence, it is seen that they have a predisposition to technology, their ability to use it in daily life, and their interests. For this reason, it is seen that technology-based applications can be used to help students learn medication applications, which are an important component of care, more willingly, permanently and effectively. Technology and mobile applications; It is a learning method that affects all cognitive, tactile, visual and kinesthetic areas. Use of technology in education; Developing independent learning skills, broadening one's views, and increasing active learning make it suitable for presenting different types of learning strategies together.

Nowadays, reasons such as the high number of students studying in nursing education programs, the insufficient number of faculty members, the increasing amount of scientific knowledge specific to nursing, the complexity of the content, and the increasing importance of students' individual differences and abilities, lead to the use of technology in nursing education and the development of these technologies. increased the need. The majority of nursing students consist of individuals who are in the generation that uses technology and the internet from an early age, and this increases the importance of integrating new technologies into nursing education. As a result of the literature review, a mobile application for subcutaneous, intramuscular and intravenous drug administration in pediatric patients that nursing students can constantly access and correct their deficiencies whenever they want has not been found. It is planned to examine the effect of the mobile application developed with the planned project on the knowledge and skill level of intravenous, intramuscular and subcutaneous drug applications, which are among the pediatric drug applications that are frequently mistaken in the literature. It is thought that with this study, the quality of nursing education will increase, students' achievements will improve, medication errors in clinics will decrease and patient safety will improve.

ELIGIBILITY:
Inclusion Criteria:

* having a smart phone
* with internet access
* agreeing to participate in the research
* completing all tabs of the mobile app

Exclusion Criteria:

* I have previously taken courses, courses, etc. on pharmaceutical applications. participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Knowledge test | through study completion-an average of 1 week
  The knowledge test developed to evaluate students' knowledge of subcutaneous, intramuscular and intravenous drug preparation and administration consists of 15 open-ended questions. The minimum values: 0 and maximum values:75. Higher scores mean a better.
Skills assessment checklist | through study completion-an average of 1 week
  It was developed to evaluate students' subcutaneous, intramuscular and intravenous drug preparation and administration skills within the scope of the Child Health and Diseases Nursing course. Checklists are used for the implementation of the course. The minimum values: 0 and maximum values:100. Higher scores mean a better.

CONTACTS AND LOCATIONS:
Overall Officials: Rukiye Çelik, Study Director — Gazi University
Locations (1):
- Gazi University, Çankaya, Ankara, Turkey (Türkiye)